CLINICAL TRIAL: NCT03973190
Title: Evaluation of Bone Quality and Primary and Secondary Stability of Implants Installed in Alveolar Regeneration Area by Three Different Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Bruno Salles Sotto-Maior, Principal investigator, Federal University of Juiz de Fora
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 51514715.9.0000.5147
Record Dates: First submitted 2019-05-27; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Alveolar Osseous Loss

STUDY DESIGN:
Intervention Model Description: Group RET: Closure of the alveolus by first intention through palatal flap sliding according to the technique of Khoury et al. (2000).
  SBC Group: Fill bone alveolus with Bone Ceramic® graft (Straumann AG, Basel, Switzerland) and cover it with palatal flap according to the technique of Khoury et al. (2000).
  PRO Group: Alveolus sealing by a temporary ovoid pony of acrylic resin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RET Group (Placebo Comparator): Closure of the alveolus by first intention through palatal flap sliding according to the technique of Khoury et al. (2000).
  Interventions: Procedure: Immediate alveolar regeneration after exodontia; Procedure: installation of dental implant and collection of biological material; Device: ISQ analysis
- SBC Group (Active Comparator): Fill bone alveolus with Bone Ceramic® graft (Straumann AG, Basel, Switzerland) and cover it with palatal flap according to the technique of Khoury et al. (2000).
  Interventions: Procedure: Immediate alveolar regeneration after exodontia; Procedure: installation of dental implant and collection of biological material; Device: ISQ analysis
- PRO Group (Active Comparator): Alveolus sealing by a temporary ovoid pony of acrylic resin.
  Interventions: Procedure: Immediate alveolar regeneration after exodontia; Procedure: installation of dental implant and collection of biological material; Device: ISQ analysis

INTERVENTIONS:
Procedure: Immediate alveolar regeneration after exodontia — The extractions will be performed under local anesthesia, without making a mucoperiosteal flap, making an intraassucular incision and using appropriate periotomes, elevators and forcépes, minimizing the surgical trauma of surrounding tissues. Thorough curettage of the alveolus will be performed at the time of extraction to ensure removal of all granulation tissue and stimulate bleeding from the bone base, to form blood clot and promote healing. The sutures will be removed after 7 days of surgery, except for patients in group 3, in which sutures will not be made.
  Other Names: alveolar regeneration and implant insertion
Procedure: installation of dental implant and collection of biological material — The material was collected for histological analysis, extracted with trephine drill of 2.0 mm in diameter. Samples were removed before the incision. A linear incision was then made on the alveolar ridge in the region and flap detachment. The initial insertion of the implant was performed using the contra-angle at 30 rpm, the final insertion of the implant was performed with manual torque wrench, where the insertion torque was measured and the value was tabulated, not exceeding 60 N. cm. The component was installed with a maximum torque of 20 N and SmartPeg® (Integration Diagnostics AB, Göteborg, Sweden) was adapted. The prosthetic component was installed with a maximum torque of 20 N and SmartPeg® (Integration Diagnostics AB, Göteborg, Sweden) was adapted. the tabulated values and the incision was sutured.
  Other Names: installation of dental implant and collection of osseous and gingival tissue
Device: ISQ analysis — The prosthetic component already installed. On it is adapted the SmartPeg® (Integration Diagnostics AB, Göteborg, Sweden). According to the manufacturer, the device generates a series of signals with different frequencies in Hertz (Hz) and these values are immediately converted to ISQ (Implantation Stability Coefficient), providing fast and accurate monitoring. The calibration is performed on the buccal and palatal surfaces of the intermediaries, that is, each implant was submitted to 2 readings. The readings were captured and tabulated for further analysis. were repeated at intervals of 7 to 10 days, 30 days and 60 days, for evaluation of SSI in the period of osseointegration. With the objective of not subjecting the implant to torque and torque during this period and to avoid interfering with the osseointegration process, the micro-pillars were covered with the micro-pillar protection screws with digital pressure only.
  Other Names: ISQ measurement

SUMMARY:
The objective of this randomized controlled clinical study was to compare bone quality between three different alveolar ridge preservation methods, also with the evaluation of primary and secondary dental implant stabilities at these sites.

DETAILED DESCRIPTION:
In the present study will be collected 24 patients, with indication of extraction of premolars or upper incisors. All participants will sign a Free and Informed Consent Form (TCLE), agreeing to participate voluntarily in this research.

Patients were randomly allocated into three groups according to the following treatments:

Group RET: Closure of the alveolus by first intention through palatal flap sliding according to the technique of Khoury.

SBC Group: Fill bone alveolus with Bone Ceramic® graft (Straumann AG, Basel, Switzerland) and cover it with palatal flap according to the technique of Khoury.

PRO Group: Alveolus sealing by a temporary ovoid pony of acrylic resin.

All patients will be prescribed the use of amoxicillin 2G, dexamethasone 4 mg and dipyrone sodium 500 mg one hour before the surgical procedure. After intra- and extraoral antisepsis with 0.12% and 2% chlorhexidine respectively, the sterile surgical fields were placed. Local anesthesia was obtained with lidocaine 2% epinephrine 1: 100,000.

With the aid of a surgical guide will be collected material for histological analysis, removed using trephine drill with 2.0 mm diameter. Samples will be removed before the incision, to be defined through the presence of gingival tissue the most coronal part of the sample. They will be placed immersed in a container with 10% formalin solution.

Then a linear incision will be made on the alveolar ridge in the region and detachment of the flap. The implants and components to be used are from Neodent® (Curitiba, PR, Brazil). The diameters used were standardized in 3.5 x 11.5 mm or 3.5 x 8 mm, depending on the remaining height of the collar. The milling and insertion system of the implants will follow the protocol recommended by the manufacturer. The drill rotation of the drills does not exceed 800 rpm, as recommended for Type III and IV bones.

The initial insertion of the implant will occur with the use of the contra-angle regulated at 30 rpm, the final insertion of the implant will be performed using a manual torque wrench, to measure the insertion torque and the registered value, preferably not exceeding 60 N.cm.The prosthetic component should be installed immediately after installation with an implant with a maximum torque of 20 N and on it adapted the SmartPeg® (Integration Diagnostics AB, Göteborg, Sweden). According to the manufacturer, the device generates a series of signals with different frequencies in Hertz (Hz) and these values are immediately converted to ISQ (Implantation Stability Coefficient), providing fast and accurate monitoring. The ISQ linear scale ranges from 1 to 100, with high ISQ values assuming high quality bone implant anchors. The calibration will be performed on the buccal and palatal surfaces of the intermediaries, that is, each implant submitted to 2 readings. The readings will be captured and recorded for further analysis.

Patients who do not achieve a minimum insertion torque of 30 N will have the micro-abutments removed, the implant cover screw installed, and sutured. In these patients, they will not have the values of SSI in the period of osseointegration of the implants. Implants that presented insertion torque equal to or greater than 30 N were to be maintained with the prosthetic components in position to have the repeated evaluations at intervals of 7 to 10 days, 30 days and 60 days, for evaluation of SSI in the period of osseointegration. With the objective of not subjecting the implant to torque and torque during this period and to avoid interfering with the osseointegration process, the micro-piers will be covered with the micro-pillar protection screws with digital pressure only, and the incision will be sutured.

Patients will receive guidance regarding postoperative care. It will be prescribed amoxicillin 500mg every eight hours for seven days, nimesulide 100mg twelve in twelve hours for three days, dipyrone sodium 500mg in case of pain and mouthwashes with chlorhexidine 0.12% of twelve in twelve hours until the removal of the sutures.After the surgical procedure, periapical radiographs of the operated region will be performed to check the position of the implants.

The microCT examination of each bone sample will be performed by the Skyscan® micrograph 1272 (Skyscan, Antwerp, Belgium) to analyze the bone microarchitecture of each location from which the implants were installed. After the analysis the samples will be subimeted to immunohistochemical tests.

ELIGIBILITY:
Inclusion Criteria:

* Extraction of premolars
* Canines or incisors
* Having two adjacent teet
* Due to root fracture
* Extensive cavities that do not allow restorative treatment and / or unfavorable -endodontic prognosis
* Systemically healthy

Exclusion Criteria:

* Patients who use any drug that influences bone metabolism
* Patients with a history of head and neck radiotherapy
* Patients undergoing chemotherapy for the treatment of malignant tumors at the time of the study
* Patients with severely resorbed alveoli
* Smokers
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-06-25 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
ISQ analysis | up to the conclusion of the study, an average of 2 years
  result and closer Immediate / at the time of surgery (values from 0-100) where 0 is closest if zero is worse the to 100 the better.After 7 days (values from 0-100) where 0 is the closest to zero the result is worse and closer to 100 the better.
  After 7 days (values from 0-100) where 0 is the closest to zero the result is worse and closer to 100 the better.
  After 30 days (values from 0-100) where 0 is the closest to zero the result is worse and closer to 100 the better.
  After 60 days (values from 0-100) where 0 is the closest to zero the result is worse and closer to 100 the better.

CONTACTS AND LOCATIONS:
Locations (1):
- Programa de Pós-graduação em Odontologia Faculdade de Odontologia - UFJF, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
will be necessary the contact with the researcher
Supporting Information: SAP, ICF, CSR
Time Frame: to be defined
Access Criteria: to be defined

REFERENCES:
- [Background] Acil Y, Sievers J, Gulses A, Ayna M, Wiltfang J, Terheyden H. Correlation between resonance frequency, insertion torque and bone-implant contact in self-cutting threaded implants. Odontology. 2017 Jul;105(3):347-353. doi: 10.1007/s10266-016-0265-2. Epub 2016 Aug 18. PMID 27538921
- [Background] Antunes AA, Grossi-Oliveira GA, Martins-Neto EC, Almeida AL, Salata LA. Treatment of circumferential defects with osseoconductive xenografts of different porosities: a histological, histometric, resonance frequency analysis, and micro-CT study in dogs. Clin Implant Dent Relat Res. 2015 Jan;17 Suppl 1:e202-20. doi: 10.1111/cid.12181. Epub 2013 Nov 28. PMID 24283568
- [Background] Araujo M, Linder E, Lindhe J. Effect of a xenograft on early bone formation in extraction sockets: an experimental study in dog. Clin Oral Implants Res. 2009 Jan;20(1):1-6. doi: 10.1111/j.1600-0501.2008.01606.x. PMID 19126101
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Background] Artzi Z, Tal H, Dayan D. Porous bovine bone mineral in healing of human extraction sockets. Part 1: histomorphometric evaluations at 9 months. J Periodontol. 2000 Jun;71(6):1015-23. doi: 10.1902/jop.2000.71.6.1015. PMID 10914806
- [Background] Barone A, Borgia V, Covani U, Ricci M, Piattelli A, Iezzi G. Flap versus flapless procedure for ridge preservation in alveolar extraction sockets: a histological evaluation in a randomized clinical trial. Clin Oral Implants Res. 2015 Jul;26(7):806-13. doi: 10.1111/clr.12358. Epub 2014 Mar 1. PMID 24580835
- [Background] Bataineh AB, Al-Dakes AM. The influence of length of implant on primary stability: An in vitro study using resonance frequency analysis. J Clin Exp Dent. 2017 Jan 1;9(1):e1-e6. doi: 10.4317/jced.53302. eCollection 2017 Jan. PMID 28149455
- [Background] Baumer D, Zuhr O, Rebele S, Hurzeler M. Socket Shield Technique for immediate implant placement - clinical, radiographic and volumetric data after 5 years. Clin Oral Implants Res. 2017 Nov;28(11):1450-1458. doi: 10.1111/clr.13012. Epub 2017 Mar 23. PMID 28333394
- [Background] Becker W, Sennerby L, Bedrossian E, Becker BE, Lucchini JP. Implant stability measurements for implants placed at the time of extraction: a cohort, prospective clinical trial. J Periodontol. 2005 Mar;76(3):391-7. doi: 10.1902/jop.2005.76.3.391. PMID 15857073
- [Background] Bornstein MM, Hart CN, Halbritter SA, Morton D, Buser D. Early loading of nonsubmerged titanium implants with a chemically modified sand-blasted and acid-etched surface: 6-month results of a prospective case series study in the posterior mandible focusing on peri-implant crestal bone changes and implant stability quotient (ISQ) values. Clin Implant Dent Relat Res. 2009 Dec;11(4):338-47. doi: 10.1111/j.1708-8208.2009.00148.x. Epub 2009 Apr 23. PMID 19438966
- [Background] Bornstein MM, Valderrama P, Jones AA, Wilson TG, Seibl R, Cochran DL. Bone apposition around two different sandblasted and acid-etched titanium implant surfaces: a histomorphometric study in canine mandibles. Clin Oral Implants Res. 2008 Mar;19(3):233-41. doi: 10.1111/j.1600-0501.2007.01473.x. Epub 2008 Jan 3. PMID 18177427
- [Background] Bouwman WF, Bravenboer N, Frenken JWFH, Ten Bruggenkate CM, Schulten EAJM. The use of a biphasic calcium phosphate in a maxillary sinus floor elevation procedure: a clinical, radiological, histological, and histomorphometric evaluation with 9- and 12-month healing times. Int J Implant Dent. 2017 Dec;3(1):34. doi: 10.1186/s40729-017-0099-x. Epub 2017 Jul 25. PMID 28741276
- [Background] Buser D, Broggini N, Wieland M, Schenk RK, Denzer AJ, Cochran DL, Hoffmann B, Lussi A, Steinemann SG. Enhanced bone apposition to a chemically modified SLA titanium surface. J Dent Res. 2004 Jul;83(7):529-33. doi: 10.1177/154405910408300704. PMID 15218041
- [Background] Santamaria-Arrieta G, Brizuela-Velasco A, Fernandez-Gonzalez FJ, Chavarri-Prado D, Chento-Valiente Y, Solaberrieta E, Dieguez-Pereira M, Vega JA, Yurrebaso-Asua J. Biomechanical evaluation of oversized drilling technique on primary implant stability measured by insertion torque and resonance frequency analysis. J Clin Exp Dent. 2016 Jul 1;8(3):e307-11. doi: 10.4317/jced.52873. eCollection 2016 Jul. PMID 27398182
- [Background] Valdec S, Pasic P, Soltermann A, Thoma D, Stadlinger B, Rucker M. Alveolar ridge preservation with autologous particulated dentin-a case series. Int J Implant Dent. 2017 Dec;3(1):12. doi: 10.1186/s40729-017-0071-9. Epub 2017 Mar 30. PMID 28361377
- [Background] Morjaria KR, Wilson R, Palmer RM. Bone healing after tooth extraction with or without an intervention: a systematic review of randomized controlled trials. Clin Implant Dent Relat Res. 2014 Feb;16(1):1-20. doi: 10.1111/j.1708-8208.2012.00450.x. Epub 2012 Mar 8. PMID 22405099
- [Background] Qabbani AA, Razak NHA, Kawas SA, Sheikh Abdul Hamid S, Wahbi S, Samsudin AR. The Efficacy of Immediate Implant Placement in Extraction Sockets for Alveolar Bone Preservation: A Clinical Evaluation Using Three-Dimensional Cone Beam Computerized Tomography and Resonance Frequency Analysis Value. J Craniofac Surg. 2017 Jun;28(4):e318-e325. doi: 10.1097/SCS.0000000000003569. PMID 28230596
- [Background] Park SH, Park KS, Cho SA. Comparison of removal torques of SLActive(R) implant and blasted, laser-treated titanium implant in rabbit tibia bone healed with concentrated growth factor application. J Adv Prosthodont. 2016 Apr;8(2):110-5. doi: 10.4047/jap.2016.8.2.110. Epub 2016 Apr 21. PMID 27141254
- [Background] Mello CC, Lemos CAA, Verri FR, Dos Santos DM, Goiato MC, Pellizzer EP. Immediate implant placement into fresh extraction sockets versus delayed implants into healed sockets: A systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2017 Sep;46(9):1162-1177. doi: 10.1016/j.ijom.2017.03.016. Epub 2017 May 3. PMID 28478869